CLINICAL TRIAL: NCT06074887
Title: The Effect of Transtheoretical Model-based Cardiac Rehabilitation Training on Self-care, Quality of Life, and Self-efficacy in Patients With Heart Failure
Brief Title: The Effect of Model-based Cardiac Rehabilitation on Self-care, Quality of Life, and Self-efficacy in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hakan ÇELİK, Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2023-12974
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2023-10

CONDITIONS: Self Care
Keywords: Transtheoretical Model; Cardiac Rehabilitation; Heart Failure; Self Care; Quality of Life; Self Efficacy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- İntervention group (Experimental): Transtheoretical model-based cardiac rehabilitation group
  Interventions: Behavioral: transtheoretical model-based intervention
- Control group (No Intervention): No intervention group

INTERVENTIONS:
Behavioral: transtheoretical model-based intervention — Pretest data are collected for patients in the intervention group in a face-to-face interview in the hospital setting.
  The training prepared according to the behavior change phase will be conducted one week later in the patients' home environment and the required data will be collected.
  In the fourth week of the research, the patient is visited at home, the training prepared according to the behavior change phase is performed at the patient's home, and the required data will be collected.
  In the eighth week of the research, the patient is visited at home, the training prepared according to the behavior change phase is performed at the patient's home, and the required data will be collected.
  In the twelfth week of the study, post-tests will be collected in the hospital.
  Arms: İntervention group

SUMMARY:
The main reason why heart failure (HF) is an important public health problem is that the incidence of HF is increasing and mortality rates remain unchanged despite the decline in the incidence of coronary artery disease. The ageing population and improved medical care services are the main factors supporting this increase. In the guidelines, education and rehabilitation are recommended for symptomatic HF patients with the highest level of evidence and recommendation (Class 1A) and considered as an integral part of HF treatment. The aim of this study was to investigate the effect of Transtheoretical Model-based cardiac rehabilitation training on self-care, quality of life and self-efficacy levels of HF patients. The study was conducted with a parallel-group, randomised controlled experimental design with pre-test and post-test measurements. Thirty-two experimental and 31 control patients, randomly assigned according to inclusion and exclusion criteria, were followed up at home for 12 weeks. Transtheoretical Model (TTM)-based CR training was applied to the intervention group through home visits. Data were collected through socio-demographic information form, behaviour change stage diagnostic form, Minnesota Living with Heart Failure Scale, European Heart Failure Self-Care Behaviour Scale, General Self-Efficacy Scale, home visit follow-up chart, patient follow-up form, telephone counselling follow-up chart and general condition assessment form. Number, percentage, mean and standard deviation were used for descriptive statistics; independent and dependent sample t-test, repeated measures ANOVA test, Chi-Square test, Fisher's Exact test, Fisher-Freeman-Halton Exact test, Wilcoxon Signed Ranks test, Mann-Whitney U test and Friedman test were used for comparative analyses. The findings showed that the TTM-based KR programme had a statistically significant effect on increasing the quality of life, self-efficacy and self-care levels and improving the clinical parameters of the patients in the intervention group. Improvement was observed in the NYHA classification of the patients in the intervention group and 96.9% of them were determined to have passed to the 'movement' stage of TTM. It is recommended that home-based CR programmes should be disseminated and health professionals should be trained in TTM-based interventions to improve the general condition and clinical parameters of HF patients. It is also recommended to investigate the effectiveness of TTM-based training programmes in different patient groups and to evaluate their long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of HF, being in classes 1, 2 and 3 according to NYHA functional classification and having an ejection fraction >30, being over 40 years of age, living within the borders of Adana province, having a telephone, and volunteering to participate in the study.

Exclusion Criteria:

* Not being able to participate in practices regularly, having CR contraindications (Hypertrophic HF, aortic stenosis, angina pectoris, oncological diagnosis, advanced COPD, having received dialysis treatment, having had an MI for less than 6 months, pregnancy and obesity), and being actively enrolled in the CR program.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
European Heart Failure Self-Care Behavior Scale | 12 weeks
  Turkish validity and reliability study of this measurement tool, which measures the self-care behaviors of HF patients, by Baydemir et al. (2013). This scale consists of 12 items, 4 sub-dimensions and a 5-point Likert structure. A low score obtained from the scale indicates high self-care behavior

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire | 12 weeks
  The Turkish validity and reliability study of this scale, which measures the quality of life of HF patients, was conducted by Özdemir (2009). This scale consists of 21 items, 2 sub-dimensions and a 6-point structure. A low score obtained from the scale indicates a high quality of life.
General Self-Efficacy Scale | 12 weeks
  The Turkish validity and reliability study of this measurement tool, which measures the self-efficacy level of individuals, was conducted by Aypay (2010). This scale consists of 10 items, 1 sub-dimension and a 4-point Likert structure. A low score obtained from the scale indicates that the general self-efficacy level is low.

CONTACTS AND LOCATIONS:
Locations (1):
- HOSPİTAL, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Background] Chouinard MC, Robichaud-Ekstrand S. Predictive value of the transtheoretical model to smoking cessation in hospitalized patients with cardiovascular disease. Eur J Cardiovasc Prev Rehabil. 2007 Feb;14(1):51-8. doi: 10.1097/HJR.0b013e328014027b. PMID 17301627
- [Background] Degertekin M, Erol C, Ergene O, Tokgozoglu L, Aksoy M, Erol MK, Eren M, Sahin M, Eroglu E, Mutlu B, Kozan O. [Heart failure prevalence and predictors in Turkey: HAPPY study]. Turk Kardiyol Dern Ars. 2012 Jun;40(4):298-308. doi: 10.5543/tkda.2012.65031. Turkish. PMID 22951845
- [Background] Gonzalez B, Lupon J, Herreros J, Urrutia A, Altimir S, Coll R, Prats M, Valle V. Patient's education by nurse: what we really do achieve? Eur J Cardiovasc Nurs. 2005 Jun;4(2):107-11. doi: 10.1016/j.ejcnurse.2005.03.006. PMID 15904880
- [Background] Li X, Yang S, Wang Y, Yang B, Zhang J. Effects of a transtheoretical model - based intervention and motivational interviewing on the management of depression in hospitalized patients with coronary heart disease: a randomized controlled trial. BMC Public Health. 2020 Mar 30;20(1):420. doi: 10.1186/s12889-020-08568-x. PMID 32228532
- [Background] Paradis V, Cossette S, Frasure-Smith N, Heppell S, Guertin MC. The efficacy of a motivational nursing intervention based on the stages of change on self-care in heart failure patients. J Cardiovasc Nurs. 2010 Mar-Apr;25(2):130-41. doi: 10.1097/JCN.0b013e3181c52497. PMID 20168193
- [Background] Zhu LX, Ho SC, Sit JW, He HG. The effects of a transtheoretical model-based exercise stage-matched intervention on exercise behavior in patients with coronary heart disease: a randomized controlled trial. Patient Educ Couns. 2014 Jun;95(3):384-92. doi: 10.1016/j.pec.2014.03.013. Epub 2014 Mar 29. PMID 24726785 (Retraction: PMID 24976395 J Adv Nurs. 2014 Oct;70(10):2414)
- [Background] Baydemir C, Ozdamar K, Unalir A. Validity of the Turkish version of the European Heart Failure Self-Care Behavior Scale. Anadolu Kardiyol Derg. 2013 Sep;13(6):573-9. doi: 10.5152/akd.2013.141. Epub 2013 May 10. PMID 23665988
- See also: Özdemir, V. A. (2009). Kronik kalp yetmezliği olan hastalarda yaşam kalitesinin değerlendirilmesi (Doctoral dissertation, Marmara Universitesi (Turkey)). — https://www.proquest.com/docview/2571088679?pq-origsite=gscholar&fromopenview=true
- See also: Aypay, A. 2010. "Öz yeterlik ölçeğinin Türkçe'ye uyarlama çalışması", İnönü Üniversitesi Eğitim Fakültesi Dergisi, 11(2), 113-131. — https://dergipark.org.tr/en/pub/inuefd/issue/8702/108659